CLINICAL TRIAL: NCT00995787
Title: A Randomized, Single-blind, Placebo-controlled, Phase I Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD1656 Compared to Placebo in T2DM Patients Treated With Metformin and Sulfonylurea
Brief Title: Safety and Tolerability of AZD1656 in Type 2 Diabetes Mellitus (T2DM) Patients Treated With Metformin and Sulfonylurea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: D1020C00026
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2010-02

CONDITIONS: Type II Diabetes Mellitus
Keywords: Type II diabetes mellitus; metformin; sulfonylurea
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — AZD1656

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD1656 (Experimental)
  Interventions: Drug: AZD1656
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1656 — Dose titration of oral suspension of AZD165 during 3 days to a tolerable dose given twice daily. Subjects will thereafter be treated with this dose twice daily for another 6 days
  Arms: AZD1656
Drug: Placebo — Dose titration of oral suspension of placebo during 3 days given twice daily. Subjects will thereafter be for another 6 days
  Arms: Placebo

SUMMARY:
The primary aim of this study is to evaluate the safety and tolerability of AZD1656 in T2DM patients treated with metformin and sulfonylurea.

ELIGIBILITY:
Inclusion Criteria:

* Male or females of non-childbearing potential
* Patients treated with a combination of Metformin and SU (glyburide, glimepiride, glibenclamide, glipizide or gliclazide) in stable doses for at least 2 months prior to enrolment visit
* Patients should have FPG in the range of 6,0 to 14 mmol/L (108 to 250 mg/dL) at enrolment and on the morning of randomisation

Exclusion Criteria:

* History of ischemic heart disease, symptomatic heart failure, stroke, transitory ischemic attack or symptomatic peripheral vascular disease
* Impaired renal function in terms of GFR<60 ml/min
* Use of insulin, glitazones, gemfibrozil, warfarin, amiodarone within 3 months prior to enrolment (screening) and use of potent CYP450 inhibitors, e.g., ketoconazole within 14 days before randomisation

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Safety variables (AE, BP, pulse, plasma glucose, laboratory variables, weight and ECG | AE will be collected from the time for randomisation until follow-up visit. Safety variables and vital signs will be measured at the pre-entry, during study days -2 to 10 and at the follow-up visit.

SECONDARY OUTCOMES:
Pharmacokinetic variables: (Area under the plasma concentration vs. time curve (AUC), maximum plasma concentration (Cmax), time to reach maximum plasma concentration (tmax), terminal elimination half-life (t½) and apparent oral clearance (CL/F) | Blood samples for analysis of plasma concentrations of AZD1656 will be collected on study days 6 and 9. The samples for analysis of glipizide will be collected on study days -1 and 6.
Pharmacodynamic variables: 24 h plasma glucose, Insulin | Samples for 24-hour plasma glucose and insulin will be collected on study days -1, 6 and 9.

CONTACTS AND LOCATIONS:
Overall Officials: Klas Malmberg, MD, PhD, Study Director — AstraZeneca R&D Mölndal, SE-431 83 Mölndal, Sweden; Marcus Dr. Marcus Hompesch, Dr, Principal Investigator — Profil Institute for Clinical Research Inc.855 3rd Avenue, Suite 4400Chula VistaCA 91911, USA
Locations (1):
- Research Site, San Diego, California, United States